CLINICAL TRIAL: NCT03680521
Title: A Phase 2 Study of Sitravatinib in Combination With Nivolumab in Patients Undergoing Nephrectomy for Locally-Advanced Clear Cell Renal Cell Carcinoma
Brief Title: Neoadjuvant Sitravatinib in Combination With Nivolumab in Patients With Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 516-002
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: ccRCC; MGCD516; Antineoplastic Agents; Immunologic factors; nivolumab; Tyrosine Kinase Inhibitor; VEGFR; TAM RTKs; PD-1; PD-L1
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sitravatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sitravatinib and nivolumab (Experimental): Sitravatinib oral capsule administered daily 2 weeks alone then in combination with nivolumab administered as 240 mg IV every 2 weeks. Total treatment duration: 6-8 weeks prior to planned nephrectomy.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Sitravatinib — Sitravatinib oral capsule administered daily for 6-8 weeks in segments 1 and 2.
Drug: Nivolumab — Nivolumab administered as 240 mg IV every 2 weeks for 4-6 weeks in segment 2.

SUMMARY:
The study will evaluate the clinical activity of sitravatinib in combination with nivolumab in patients with locally-advanced clear cell renal cell carcinoma (ccRCC) in the neoadjuvant setting prior to nephrectomy.

DETAILED DESCRIPTION:
Sitravatinib is a receptor tyrosine kinase inhibitor (TKI) that targets multiple closely related receptor tyrosine kinase pathways including VEGFR, PDGFR, c-KIT, MET, and the TAM family of receptors (TYRO3, AXL, and MER). Nivolumab is a monoclonal antibody directed against PD-1 and blocks the interaction between PD-1 and its ligands, thereby releasing PD-1-mediated inhibition of T-cell proliferation (including cytotoxic CD8+ T-cells) and cytokine production. Together, sitravatinib and nivolumab may cooperate to elicit greater anti-tumor activity than either agent alone, as sitravatinib is predicted to enhance several steps in the cancer immunity cycle that may augment the efficacy of nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging results consistent with locally-advanced RCC
2. Candidate for partial or complete nephrectomy as part of treatment plan.
3. Measurable disease per RECIST version 1.1.
4. ECOG performance status 0 or 1.
5. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Prior systemic anti-tumor treatment for RCC.
2. Patients who are receiving any other investigational agents.
3. Clinical status indicating that immediate surgery (within 6 weeks) is warranted regardless of whether neoadjuvant therapy is to be administered, as assessed by the treating surgeon.
4. Inability to undergo baseline tumor biopsy.
5. Active or prior documented autoimmune or immunocompromising conditions.
6. Uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the participants completed screening, participants underwent an initial diagnostic tumor biopsy of their renal lesion. Out of the 25 participants enrolled, 5 participants did not receive treatment per protocol. The reasons were ineligible histology (3), disallowed concomitant treatment (1), and patient noncompliance (1).
Groups:
- Sitravatinib 120 mg: Participants received sitravatinib orally, once a day, at a dose of 120 mg for 2 weeks (segment 1). Then, the participants continued to receive sitravatinib in combination with nivolumab 240 mg administered as an intravenous (IV) infusion every 2 weeks, for a maximum of 6 additional weeks (segment 2).
- Sitravatinib 80 mg: Participants received sitravatinib orally, once a day, at a dose of 80 mg for 2 weeks (segment 1). Then, the participants continued to receive sitravatinib in combination with nivolumab 240 mg administered as an intravenous (IV) infusion every 2 weeks, for a maximum of 6 additional weeks (segment 2).
Period: Overall Study
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Started | 7 | 13
Completed | 7 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of either sitravatinib or nivolumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (6.19) | 56.7 (12.70) | 59.1 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 12 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — EGOG performance status was measured on a 6 point scale to assess participant's performance status.
  0: Fully active, able to carry on all pre-disease performance without restriction
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 7 | 12 | 19
    1 | 0 | 1 | 1
Clinical TNM Staging at Diagnosis [Count of Participants; unit: Participants] — T = Size of original tumour, classed from T0 to T4; N = Degree of spread to lymph nodes classed from N0 to N3; M = Presence of distant metastasis classed as M0 to M1. X denotes uncertainty in assigning a given category (T, N, or M) when all reasonable clinical or pathologic maneuvers have been used in staging.
  Participants
    T2bN0M0 | 1 | 0 | 1
    T3N0M0 | 0 | 1 | 1
    T3N0M1 | 0 | 1 | 1
    T3NXM0 | 0 | 1 | 1
    T3aN0M0 | 6 | 2 | 8
    T3aNXM0 | 0 | 7 | 7
    T3aNXM1 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Point in Time Objective Response (Either Complete or Partial Response [CR or PR]) Prior to Surgery
Description: Objective response is defined as the percent of participants documented by investigator assessment to have Complete Response (CR) or Partial Response (PR) in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). CR is defined as complete disappearance of all baseline target and non-target lesions with the exception of nodal disease; PR is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: Clinical activity evaluable population: All participants who 1) had measurable disease (per RECIST 1.1) at baseline, 2) received at least one dose of both sitravatinib and nivolumab, 3) had their onstudy disease assessment prior to surgery, and 4) underwent surgery and were deemed disease-free (i.e. non-metastatic) after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 6 | 11
Participants | 2 | 0

2. Primary Outcome: Point in Time Objective Response Prior to Surgery
Description: Number and percentage of participants who experienced a response prior to surgery in accordance with RECIST 1.1.
  * CR is defined as complete disappearance of all baseline target and non-target lesions with the exception of nodal disease;
  * PR is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions;
  * Stable Disease (SD) is concluded when the single point in time response does not qualify for CR, PR or Progressive Disease (PD);
  * PD is defined as a 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing nontarget lesions.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 6 | 11
Participants
  Preoperative timepoint response: CR | 0 | 0
  Preoperative timepoint response: PR | 2 | 0
  Preoperative timepoint response: SD | 4 | 11
  Preoperative timepoint response: PD | 0 | 0

3. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs occured after the first dose of any study treatment or any preexisting condition that increased in severity after the first dose of study treatment and prior to 28 days after last dose of study drug or surgery, whichever occurred last.
  TEAEs were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Day 1 until 28 days after last dose of study drug or surgery, whichever occurred last (up to a maximum of 13 weeks)
Population: Safety population: all participants who received at least 1 dose of either sitravatinib or nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 7 | 13
Participants | 7 | 13

4. Secondary Outcome: Blood Plasma Concentrations of Sitravatinib
Description: The blood plasma concentrations of sitravatinib were determined using blood samples. Blood samples for analysis of blood plasma concentrations of sitravatinib were taken after scheduled vital signs and triplicate electrocardiogram assessments.
Time Frame: Day 1 (pre-dose, and 30 minutes and 4 hours post-dose), Day 15 (pre-dose) and Day 43 (pre-dose)
Population: Pharmacokinetics (PK) evaluable population: all participants who received treatment with sitravatinib and had non-missing concentration-time data. Concentration was assessed by actual dose associated with each time-point. One participant was randomized to sitravatinib 120 mg arm, but received sitravatinib 60 mg at Day 43.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PK Population: Sitravatinib 120 mg: PK assessments were assessed based on the actual dose associated with the visit. The PK assessment was associated with a daily dose of 120 mg of sitravatinib orally.
- PK Population: Sitravatinib 80 mg: PK assessments were assessed based on the actual dose associated with the visit. The PK assessment was associated with a daily dose of 80 mg of sitravatinib orally.
- PK Population: Sitravatinib 60 mg: PK assessments were assessed based on the actual dose associated with the visit. The PK assessment was associated with a daily dose of 60 mg of sitravatinib orally. This participant was randomized to sitravatinib 120 mg arm, but received sitravatinib 60 mg at Day 43.
Arm/Group | PK Population: Sitravatinib 120 mg | PK Population: Sitravatinib 80 mg | PK Population: Sitravatinib 60 mg
Number analyzed (Participants) | 7 | 13 | 1
ng/mL
  Day 1 (pre-dose): number analyzed (Participants) | 7 | 13 | 0
  Day 1 (pre-dose) | 0.0 (0.00) | 0.6 (2.27) |
  Day 1 (30 mins post-dose): number analyzed (Participants) | 7 | 13 | 0
  Day 1 (30 mins post-dose) | 2.9 (2.12) | 1.0 (1.17) |
  Day 1 (4 hours post-dose): number analyzed (Participants) | 7 | 13 | 0
  Day 1 (4 hours post-dose) | 17.0 (10.38) | 13.7 (10.60) |
  Day 15 (pre-dose): number analyzed (Participants) | 3 | 10 | 0
  Day 15 (pre-dose) | 87.7 (9.62) | 63.3 (42.36) |
  Day 43 (pre-dose): number analyzed (Participants) | 5 | 5 | 1
  Day 43 (pre-dose) | 75.0 (23.74) | 53.7 (32.88) | 66.5 (NA) — Only 1 participant received 60 mg, so standard deviation (SD) could not be calculated.

5. Secondary Outcome: Time to Surgery
Description: Time to surgery was defined as the number of calendar days between Day 1 and the planned nephrectomy.
Time Frame: Day 1 up to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 6 | 11
days
  Time to Surgery | 56.5 [46.0 to 61.0] | 50.0 [46.0 to 55.0]
  Delays in Surgery | 1.0 [1 to 4] | 1.0 [1 to 39]

6. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS was defined as the time from date of surgery to disease recurrence or death whichever occurred first.
Time Frame: Up to 3 years after surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 6 | 11
months | NA [32.13 to NA] — Median and upper confidence interval data could not be analyzed because too few participants experienced an event of disease recurrence or death. | NA [18.56 to NA] — Median and upper confidence interval data could not be analyzed because too few participants experienced an event of disease recurrence or death.

7. Secondary Outcome: Percentage Change From Baseline in Programmed Death Ligand 1 (PD-L1) Expression in the Tumor
Description: Tumor tissue was collected from study biopsies and surgical samples. Tumor tissue was used to assess the mean PD-L1 expression in the tumor via immunohistochemistry and/or immunofluorescence.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: Pharmacodynamic evaluable population: all participants who received at least 1 dose of sitravatinib or nivolumab for whom sufficient pharmacodynamic data were available for analysis of the endpoint.
Measure: Mean (Standard Deviation); unit: percentage change in PD-L1 expression
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 5 | 8
percentage change in PD-L1 expression | 1.6 (2.07) | 2.5 (7.07)

8. Secondary Outcome: Change From Baseline in Myeloid-derived Suppressor Cells (MDSCs) in the Tumor
Description: Tumor tissue was collected from study biopsies and surgical samples, and was used to assess mean MDSCs using immunohistochemistry.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 2 | 3
cells/mm^2 | 34.5 (72.41) | -55.1 (151.11)

9. Secondary Outcome: Change From Baseline in Regulatory T-cells (Tregs) in the Tumor
Description: Tumor tissue was collected from study biopsies and surgical samples, and was used to assess mean Tregs using immunohistochemistry.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 2 | 3
cells/mm^2 | -24.1 (45.86) | 49.6 (43.62)

10. Secondary Outcome: Change From Baseline in CD4+ T-cells in the Tumor
Description: Tumor tissue was collected from study biopsies and surgical samples, and was used to assess mean CD4+ T-cells using immunohistochemistry.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 2 | 3
cells/mm^2 | -114.1 (144.72) | 111.2 (231.86)

11. Secondary Outcome: Change From Baseline in CD8+ T-cells in the Tumor
Description: Tumor tissue was collected from study biopsies and surgical samples, and was used to assess mean CD8+ T-cells using immunohistochemistry.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 2 | 3
cells/mm^2 | -88.3 (164.13) | 30.9 (181.86)

12. Secondary Outcome: Change From Baseline in Ratio of Type 1 to Type 2 Tumor Associated Macrophages in the Tumor
Description: Tumor tissue was collected from study biopsies and surgical samples, and was used to assess mean ratio of Type 1 to Type 2 tumor associated macrophages using immunohistochemistry.
Time Frame: Baseline to date of surgery (maximum time to surgery was approximately 13 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 2 | 3
ratio | -1.9 (2.28) | -1.1 (1.15)

13. Secondary Outcome: Change From Baseline of Selected Cytokines in Peripheral Blood
Description: Cytokines measured in peripheral blood were soluble CD27 (sCD27), eotaxin, macrophage inflammatory protein 1b (MIP-1b), and soluble programmed cell death protein 1 (sPD-1).
Time Frame: Baseline to Day 43
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
Number analyzed (Participants) | 6 | 8
pg/ml
  sCD27 | -78.6 (755.97) | -30.3 (567.82)
  Eotaxin | 3.1 (12.91) | 3.4 (12.48)
  MIP-1b | 10.6 (20.33) | 1.9 (6.58)
  sPD-1 | 3.6 (19.59) | 3.8 (12.49)

ADVERSE EVENTS:
Time Frame: All cause mortality: Up to 3 years after surgery (maximum time to surgery was approximately 13 weeks); serious and other adverse events: Day 1 until 28 days after last dose of study drug or surgery, whichever occurred last (up to a maximum of 13 weeks)
Arm/Group | Sitravatinib 120 mg | Sitravatinib 80 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/13
Other Adverse Events (participants affected / at risk) | 7/7 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitravatinib 120 mg (N=7) | Sitravatinib 80 mg (N=13)
Atypical pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitravatinib 120 mg (N=7) | Sitravatinib 80 mg (N=13)
Hypertension (Vascular disorders) | 6 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Fatigue (General disorders) | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 6
Headache (Nervous system disorders) | 4 | 3
Alanine aminotransferase increased (Investigations) | 1 | 5
Constipation (Gastrointestinal disorders) | 3 | 3
Lipase increased (Investigations) | 3 | 3
Nausea (Gastrointestinal disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Amylase increased (Investigations) | 2 | 1
Blood thyroid stimulating hormone increased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 2
Oral dysaesthesia (Gastrointestinal disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1
Pain (General disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Thyroiditis (Endocrine disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight decreased (Investigations) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Haematocrit increased (Investigations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1
Incision site vesicles (Injury, poisoning and procedural complications) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT03680521/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03680521/SAP_001.pdf